CLINICAL TRIAL: NCT06733818
Title: The Evaluation of the Levels of Physical Function in Older Adults From the Perspective of Active Ageing
Brief Title: Physical Function From the Perspective of Active Ageing
Status: Completed | Type: Observational
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Tahir Keskin , Pt, PhD, Research Assistant, Suleyman Demirel University
Other Study IDs: SuleymanDUtahirkeskin05
Record Dates: First submitted 2024-12-10; First posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Aging; Physical Functional Performance; Physical Activity; Active Ageing
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Functional assessment of physical performance — Functional assessment of physical performance was performed with the Alusti test. This 10-question test was developed to assess physical performance in the geriatric population 13 and has been validated in Turkish 14. This test evaluates limb range of motion and muscle strength, ability to move from supine to sitting position, sitting balance, ability to stand up from sitting position, standing, walking, walking distance, ability to stand on tandem and single leg with eyes closed. The results of this test, which is scored out of 100, indicate the level of activity. 0-30, interpreted as totally dependent; 31-40, highly dependent; 41-50, moderately dependent; 51-60, slightly dependent; 61-75, good activity; 76-90, very good activity; and 91-100, excellent activity.

SUMMARY:
The aim of this study is to evaluate physical function from the perspective of active aging as well as to determine the relationship between physical activity and physical performance in the context of active aging.

This cross-sectional study was conducted with the participation of 215 (47.3%) males and 230 (52.7%) females, with a mean age of 69.09±8.59 years. Functional assessment of physical performance (Alusti), Physical Activity Scale for Elderly (PASE), and University of Jyvaskyla Active Ageing Scale (UJACAS) were employed to assess physical function and active aging levels of the elderly.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 65 years and over who scored 24 points or more on the Mini Mental State Examination (MMSE) and demonstrated an ability to comprehend the instructions provided.

Exclusion Criteria:

* Individuals who were diagnosed with a neurological disorder, had undergone surgery within the past six months, had been diagnosed with cancer, lacked the capacity for verbal communication, or had severe vision impairment were excluded from the study

Ages: 55 Years to 95 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study was conducted with individuals aged 65 and over residing in the Isparta province of Turkey. The study population comprised voluntary individuals aged 65 years and over who scored 24 points or more on the Mini Mental State Examination (MMSE) and demonstrated an ability to comprehend the instructions provided.
Sampling Method: Probability Sample
Enrollment: 455 (Actual)
Dates: Start 2024-01-04 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-09-10 (Actual)

PRIMARY OUTCOMES:
Active Ageing Scale | Up to 2 months
  Active ageing was assessed using the University of Jyvaskyla Active Ageing Scale (UJACAS), developed by Rantanen et al. 15, and validated in Turkish 1. The scale consists of 17 questions and 4 subscales developed to measure active ageing. The subscales that question the main criteria of active ageing are goals (what they want to do), functional capacity (what they can do), opportunity (perceived opportunities to do activities), and activities (what they do). Participants are asked to rate the questions on a scale from 0 (lowest) to 4 (highest) for the last 4 weeks, and scoring is done accordingly. The subscales are scored between 0-68 and the total score between 0-247, with high scores associated with high levels of active ageing.

CONTACTS AND LOCATIONS:
Locations (1):
- Suleyman Demirel University Faculty of Health Sciences Physiotherapy and Rehabilitation Department, Isparta, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Keskin T, Ergan M, Baskurt Z, Baskurt F. The evaluation of the levels of physical function in older adults from the perspective of active aging. Geriatr Nurs. 2026 Jan 23;69:103845. doi: 10.1016/j.gerinurse.2026.103845. Online ahead of print. PMID 41579661